CLINICAL TRIAL: NCT02215863
Title: Immunogenicity and Safety of 13-valent Pneumococcal Conjugate Vaccine (PCV13) and MF59-adjuvanted Influenza Vaccine (Fluad) After Concomitant Vaccination in Adults Aged ≥60 Years
Brief Title: Immunogenicity and Safety of PCV13 and Fluad in Adults Aged ≥60 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Hee Jin Cheong, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FLUPCV13
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Influenza; Streptococcus Pneumoniae
Keywords: Immunogenicity, Safety, MF59, Influenza vaccine, Pneumococcal vaccine
MeSH Terms: conditions — Influenza, Human | interventions — 13-valent pneumococcal vaccine; fluad vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PCV13 and Fluad (Active Comparator): 437 concomitant Fluad-PCV13 recipients: one dose of each vaccine administered on Day 0
  Interventions: Biological: Fluad and Prevenar13
- Fluad alone (Active Comparator): 437 Fluad recipients: one vaccine injection administered on Day 0
  Interventions: Biological: Fluad
- PCV13 alone (Active Comparator): 437 PCV13 recipients: one vaccine injection administered on Day 0
  Interventions: Biological: Prevenar13

INTERVENTIONS:
Biological: Fluad and Prevenar13
  Arms: PCV13 and Fluad
Biological: Fluad
  Arms: Fluad alone
Biological: Prevenar13
  Arms: PCV13 alone

SUMMARY:
Recent reviews have highlighted the unpredictability and complexity of immune interference when multivalent conjugate vaccines are co-administered with other pediatric vaccines. It has become evident that the likelihood of immune interference (in response to conjugated- or co-administered antigens) increases in proportional to the number of glyco-conjugates (valencies) and dosages of carrier proteins. There are many kinds of carrier proteins: tetanus toxoid (TT), diphtheria toxoid (DT), CRM197 (non-toxic variant of DT), OMP (complex outer-membrane protein mixture from Neisseria meningitidis) and non-typeable Hemophilus influenza-derived protein D. Among them, TT is a more potent inducer of T-helper immunity, but carrier-induced-epitopic suppression (dose-dependent carrier antibody and carrier B cell dominance) may occur with TT. In comparison, DT and CRM197 are weaker B-cell immunogens, but apparently trigger more T-regulatory mechanism. Recent pediatric studies of PCV13 co-administered with DTaP vaccines showed 6B GMT (geometric mean titer) to be somewhat reduced compared to the results with PCV13 alone.

Similar to children, adults frequently visit outpatient clinics to get two or more kinds of vaccines at the same time: pneumococcal vaccine, influenza vaccine, Td (diphtheria and tetanus) vaccine, HPV (human papilloma virus) vaccine, meningococcal vaccine, zoster vaccine, etc. PCV13 has limited co-administration information for adjuvanted influenza vaccine.

This study is designed to evaluate the immunogenicity and safety of PCV13 and MF59-adjuvanted influenza vaccine (Fluad) after concomitant administration in adults aged 60 years or older.

DETAILED DESCRIPTION:
This study is a multi-centered, randomized controlled clinical trial: Korea University Guro Hospital, Korea University Ansan Hospital, Hallym University Gangnam Sacred Hospital and Catholic University Medical College, St. Vincent's Hospital.

The primary objective is to evaluate the immunogenicity of Fluad after concomitant administration of Fluad and PCV13 in adults aged 60 years or more. This study is designed to demonstrate non-inferiority of sero-conversion rate after Fluad vaccination: Fluad-PCV13 co-administration group versus Fluad alone group

The secondary objective is to evaluate the immunogenicity of PCV13 after concomitant administration in adults aged 60 years or more. This study is designed to demonstrate non-inferiority of PCV13 when co-administered with Fluad compared with PCV13 alone.

This study is also designed to evaluate the safety of concomitant PCV13-Fluad administration in adults aged 60 years or more. All the participants will be followed for the duration of an expected average of 4 weeks after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥60 years who signed the informed consent

Exclusion Criteria:

* Previous pneumococcal vaccine recipients
* Egg allergy
* History of serious adverse event after vaccination,
* any acute disease or infection
* History of neurological symptoms or signs
* Impairment of immune function or immunosuppressant use
* Bleeding diathesis
* Fever (defined as axillary temperature ³38.0°C) within 3 days (prior to Visit 1)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1195 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Seroconversion rates (A/H1N1, A/H3N2, and B) | Outcome measure will be assessed at two points (baseline and 4 weeks after vaccination)
  a post-vaccination titer ≥1:40 in subjects with a pre-vaccination titer of <1:10 or a ≥4-fold titer increase in subjects with a pre-vaccination titer of ≥1:10

SECONDARY OUTCOMES:
Seroprotection rates and GMT folds (A/H1N1, A/H3N2, and B) | Outcome measure will be assessed at two points (baseline and 4 weeks after vaccination).
  * Seroprotection rate: percentage of subjects with a post-vaccination titer ≥1:40
  * GMT-fold change: GMT ratio of the post-vaccination titer to pre-vaccination titer
Opsonophagocytic assay (OPA) titers for PCV13 | Outcome measure will be assessed at two points (baseline and 4 weeks after vaccination).
  OPA geometric mean titers for 13 PCV13 serotypes with corresponding 2-sided 95% confidence intervals between groups receiving PCV 13 and then compare the results

OTHER OUTCOMES:
Frequency and duration of local and systemic adverse events | All participants will be followed until 4 weeks after vaccination)
  The safety profiles of co-administration of Fluad and PCV13 will be compared to those of single vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Jin Cheong, MD, PhD, Principal Investigator — Korea University Guro Hospital; Joon Young Song, MD, PhD, Principal Investigator — Korea University Guro Hospital
Locations (3):
- South Korea (3):
  - Korea University Ansan Hospital, Ansan
  - Hallym University Gangnam Sacred Hospita, Seoul
  - Catholic University Medical College, St. Vincent's Hospital, Suwon

REFERENCES:
- [Derived] Song JY, Cheong HJ, Hyun HJ, Seo YB, Lee J, Wie SH, Choi MJ, Choi WS, Noh JY, Yun JW, Yun JG, Kim WJ. Immunogenicity and safety of a 13-valent pneumococcal conjugate vaccine and an MF59-adjuvanted influenza vaccine after concomitant vaccination in ⩾60-year-old adults. Vaccine. 2017 Jan 5;35(2):313-320. doi: 10.1016/j.vaccine.2016.11.047. Epub 2016 Dec 3. PMID 27919632